CLINICAL TRIAL: NCT06723977
Title: The Effect of Auditory Hallucination-based Sound Simulation Application That is Listened to by Caregivers of Individuals with Schizophrenia on Their Emotional Expression and Perceived Family Burden
Brief Title: Effect of Simulation on Emotional Expression and Perceived Family Burden of Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fatma Gül SAK, Principal Investigator, PhD student, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESOGÜ-SBE-FGS-01
Record Dates: First submitted 2024-07-16; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Caregiver Burden; Expressed Emotion
Keywords: schizophrenia; perceived family burden; expressed emotion; psychiatric nursing
MeSH Terms: conditions — Schizophrenia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The study was conducted with 20 caregivers of individuals diagnosed with schizophrenia in the intervention group and 20 caregivers of individuals diagnosed with schizophrenia in the control group.
Masking Description: While written consent was obtained from the individuals included in the study, a different form was used for each group. For this reason, participants could not be blinded. In addition, since the data collection and application process had to be actively managed, researcher blinding was not possible. The randomization table was prepared by an independent statistician to avoid the possibility of bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Auditory Hallucination Based Voice Hearing Simulation application was applied to the intervention group and an information brochure was given. Auditory Hallucination Based Voice Hearing Simulation was applied only once to caregivers of individuals diagnosed with schizophrenia. The application took an average of 45 minutes.
  Interventions: Other: Auditory Hallucination Based Voice Hearing Simulation
- control group (No Intervention): The control group continued the routine practices of the clinic and was given an information brochure.

INTERVENTIONS:
Other: Auditory Hallucination Based Voice Hearing Simulation — 1. st stage: Preparation of the environment, introduction, providing information about the purpose, duration and content of the application, application of data collection tools and distribution of the information brochure were provided.
  2. nd stage: Introducing the recording devices and headphones, performing the first task simultaneously while listening to the prepared three-dimensional sound recording (watching a city promotional film and answering verbal questions about this film), performing the second task simultaneously while listening to the prepared three-dimensional voice recording (telling a story). (reading the text and answering the questions about this story text in writing) were applied.
  3. rd stage: Information about the next application time of the measurement tools was provided.
  Additional stage: Data collection tools were reapplied.
  Arms: intervention group

SUMMARY:
The aim of this study is to determine the effect of Auditory Hallucination Based Voice Hearing Simulation on the emotional expression and perceived family burden of caregivers of individuals diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Objective: The aim of this study is to determine the effect of Auditory Hallucination Based Voice Hearing Simulation on the emotional expression and perceived family burden of caregivers of individuals diagnosed with schizophrenia.

Method: This study was designed in a pre-test - post-test, randomized controlled design. The study was conducted with 20 caregivers in the intervention group and 20 caregivers of individuals diagnosed with schizophrenia in the control group. Data were collected between March 2023 and October 2023 using the Emotional Expression Scale and Perceived Family Burden Scale. Auditory Hallucination Based Voice Hearing Simulation was applied to the intervention group. This sound recording is three-dimensional. While the audio recording is played to the caregivers; Users were asked to complete two tasks, each lasting 10 minutes. The tasks were carried out under the guidance prepared by the researchers. In the control group, the routine practices of the clinic continued.

ELIGIBILITY:
Inclusion Criteria:

* Having been living with an individual diagnosed with schizophrenia for at least one year.
* Being primarily responsible for the care of the individual diagnosed with schizophrenia,
* Being between the ages of 18-65,
* Being literate,
* Speaking Turkish,
* Volunteering to participate in the study.

Exclusion Criteria:

* Having a physical disability to perform the assigned tasks,
* Having any health problem related to hearing ability,
* Having any mental illness,
* Having received 2 or more points from the General Health Questionnaire-12.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Level of Expressed Emotion Scale - LEES | one month
  The scale was developed to measure the quality of social interaction between the patient and the caregiver. The scale consists of 41 items. The maximum total score obtained from the scale is 41, and the minimum is 0. High scores from the scale indicate that the caregiver has high emotional expression.
The Perceived Family Burden Scale - PFBS | one month
  This scale, which is applied to relatives of individuals diagnosed with schizophrenia, was developed to evaluate the family burden perceived by the patient's relatives. The scale, which evaluates the patient's relative's perception of family burden in the last month, consists of 24 items and two parts, A-B. The maximum total score obtained from the scale is 108, and the minimum is 0.
  The scale does not have a cut-off point, and high scores from the scale indicate a high perceived family burden.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gül Sak, PhD Student, Principal Investigator — Diyarbakır Selahaddin Eyyubi State Hospital Community Mental Health Center
Locations (1):
- Diyarbakır Selahaddin Eyyubi State Hospital Community Mental Health Center, Diyarbakır, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A utility model application will be made for the application. Therefore, the data will not be shared.